CLINICAL TRIAL: NCT05380375
Title: Short-course Versus Very Short-course Antibiotic Treatment in Acute Exacerbations of COPD: a Meta-analysis of Double-blind Studies
Brief Title: Short-course Antibiotic Treatment in AECOPD: a Meta-analysis of Double-blind Studies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professeur, University of Monastir
Other Study IDs: Meta analysis
Record Dates: First submitted 2022-05-07; First posted 2022-05-18 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: COPD Exacerbation
Keywords: AECOPD; antibiotic treatment; meta analysis; short course; Forest plot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short-course: Group with short treatment of antibiotic of <= 5 days
- Very short-course: Group with short treatment of antibiotic of <= 3 days

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common disease worldwide and a leading cause of death and disability globally. Given that bacteria are implicated in a substantial proportion of acute exacerbation of COPD (AECOPD), antibiotics are frequently used. However, this current practice may lead to antibiotic overuse further increasing drug resistance and side effects. Although the small literature on interventions to prove the effective of short course of antibiotic, a metaanalysis of published randomised double-blind studies comparing the same antibiotics compared to a previous study is performed to determine whether a short course of antibiotic treatment is as effective as a very short course in patients with an exacerbation of COPD (EACOPD). The authors systematically searched electronic databases on the literature of controlled trials on Medline and Embase with no language, location, or time restrictions. The authors retrieved observational and controlled trials comparing different durations of the same oral antibiotic therapy in the treatment of acute exacerbations of COPD. The authors included 30 randomized, placebo-controlled trials for COPD patients. There was no statistically significant difference between shorter and longer antibiotic courses in early clinical success. In conclusion, Short-course antibiotic treatment is as effective as very short-course treatment in patients with mild to moderate exacerbations of chronic bronchitis and COPD.

ELIGIBILITY:
Inclusion Criteria:

* Studies considered eligible for inclusion were randomised trials of antibiotic intervention involving adult patients >18 years of age with a diagnosis of AECOPD.

Exclusion Criteria:

* Studies not published in the English language or with more than two or different antibiotics were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We searched on the literature of controlled trials on Medline and Embase using the following search terms: COPD, antibiotic treatment and clinical trials. We also searched the reference lists of included studies for additional studies.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-03-05 (Estimated); Study Completion 2023-05-08 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 30 days
  clinical cure at early follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Semir Nouira, Monastir, Tunisia

REFERENCES:
- [Derived] Messous S, Rekik A, Keraani L, Hamed R, Toumia M, Dhaoui R, Sekma A, Ali KBH, Sassi S, Kouraichi C, Boukef R, Bouida W, Boubaker H, Msolli MA, Nouira S. Comparative Efficacy and Safety of Short- Versus Standard-course Fluoroquinolone Treatment in Acute Exacerbations of Chronic Obstructive Pulmonary Disease: A Meta-analysis of Double-blind Studies. Clin Ther. 2025 Aug;47(8):631-637. doi: 10.1016/j.clinthera.2025.04.020. Epub 2025 May 25. PMID 40414751